CLINICAL TRIAL: NCT04590339
Title: Lateralization of the Inferior Alveolar Nerve After Repositioning of the Bone Window Versus Sticky Bone Augmentation: A Randomized Controlled Clinical Trial
Brief Title: Lateralization of the Inferior Alveolar Nerve After Repositioning of the Bone Window Versus Sticky Bone Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0010556-IORG 00088390
Record Dates: First submitted 2020-08-12; First posted 2020-10-19 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Posterior Atrophic Mandible; Inferior Alveolar Nerve; Nerve Lateralization
Keywords: inferior Alveolar nerve lateralization; neurosensory disturbance; guided surgery; Posterior atrophic mandibular ridge

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Repositioning the bone window (Active Comparator): Computer guided inferior alveolar nerve lateralization and implant placement with subsequent repositioning of the osteotomized bone window.
  Interventions: Procedure: Guided inferior Alveolar Nerve lateralization
- Augmentation using sticky bone (Active Comparator): Computer guided inferior alveolar nerve lateralization and implant placement with grafting around the implant using sticky bone
  Interventions: Procedure: Guided inferior Alveolar Nerve lateralization

INTERVENTIONS:
Procedure: Guided inferior Alveolar Nerve lateralization — Evaluating neurosensory recovery after Implant placement in posterior atrophic mandible by Guided inferior alveolar nerve lateralization technique
  Other Names: computer guided implant placement

SUMMARY:
Rehabilitation of edentulous posterior mandibular regions with severe ridge atrophy using implants is subject to anatomical, surgical, and biological difficulties. In many cases, the bone is severely atrophied that sufficiently long fixtures cannot be placed without encroaching on the inferior alveolar nerve (IAN). IANL is defined as the lateralization of inferior alveolar neurovascular bundle posterior to the mental foramen, with preservation of the incisive nerve; exposure and traction are used to deflect the IAN laterally while the implants are placed.

DETAILED DESCRIPTION:
This prospective randomized clinical trial will enroll 20 patients with posterior mandibular ridge atrophy. Ten of which will undergo computer guided nerve lateralization with subsequent implant placement and repositioning of the osteomotized bone window and ten patients will undergo computer guided nerve lateralization with subsequent implant placement and sticky bone grafting.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from unilateral posterior mandibular edentulism and having < 8 mm of bone above the mandibular canal.
* The width of the ridge should be > 4mm.
* The patient should be psychologically accepting the implant and the involved procedures.
* The patients should have adequate oral hygiene and adequate bone quality.

Exclusion Criteria:

* Any absolute contraindication for implant surgery such as uncontrolled diabetes mellitus, blood and/or bleeding disorders, serious osseous defects…etc.
* Any relevant systemic disease directly affecting bone metabolism and healing.
* Any habits that might reduce the blood flow and retard healing such as heavy smoking and alcoholism.
* A history of any grafting procedure at the designated area.
* Patient with thick cortical bone buccally and a thin neurovascular bundle.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Change in neurosensory recovery and sensation regaining over 6 months compared to normal (taken at base line) | 1 month, 3 months and 6 months
  Electrophysiological test using Mental nerve Blink reflex is done for each patient before surgery(base line), after surgery at 1 month, 3 months and 6 months.
Clinical assessment of the change in neurosensory function recovery using Static light touch detection test. | 1 week, 1 month, 3 months and 6 months
  Done at 1 week, 1 month, 3 months and 6 months postoperative.
Clinical assessment of the change in neurosensory function recovery using Brush stroke discrimination test. | 1 week, 1 month, 3 months and 6 months
  Done at 1 week, 1 month, 3 months and 6 months postoperative.
Clinical assessment of the change in neurosensory function recovery using two point discrimination test | 1 week, 1 month, 3 months and 6 months
  Done at 1 week, 1 month, 3 months and 6 months postoperative.
Clinical assessment of the change in neurosensory function recovery using pin-prick sensation test. | 1 week, 1 month, 3 months and 6 months
  Done at 1 week, 1 month, 3 months and 6 months postoperative.

SECONDARY OUTCOMES:
Implant Success rate | 3 months and 6 months
  Implant Stability using osstell device to measure the implant success at the time of implant insertion, after 3 month and at 6 month.

CONTACTS AND LOCATIONS:
Overall Officials: Dina N. Metawie, Principal Investigator — Alexandria University
Locations (1):
- Dina Metawie, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No